CLINICAL TRIAL: NCT00114088
Title: Surgical Treatments Outcomes Project for Dysfunctional Uterine Bleeding (STOP-DUB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5U01HS009506 (AHRQ)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Menorrhagia; Uterine Bleeding
Keywords: Hysterectomy,; Endometrial ablation,; Ovulatory dysfunctional uterine bleeding,; Anovulatory dysfucntional uterine bleeding,; DUB; Dysfunctional uterine bleeding
MeSH Terms: conditions — Menorrhagia; Uterine Hemorrhage; Metrorrhagia | interventions — Hysterectomy; Endometrial Ablation Techniques

INTERVENTIONS:
Procedure: hysterectomy
Procedure: endometrial ablation

SUMMARY:
STOP-DUB is a multicenter randomized clinical trial that is assessing the efficacy and effectiveness of hysterectomy versus endometrial ablation (EA) for dysfunctional uterine bleeding (DUB) in women for whom medical management has not provided relief.

DETAILED DESCRIPTION:
The Surgical Treatments Outcomes Project for Dysfunctional Uterine Bleeding (STOP-DUB) is a multicenter, randomized clinical trial that assessed the efficacy and effectiveness of hysterectomy versus endometrial ablation (EA) for dysfunctional uterine bleeding (DUB) in women for whom medical management has not provided relief. Institutional review board-approved study sites included the coordinating center, chair's office, the American College of Obstetricians and Gynecologists, and 33 clinical centers in the United States and Canada. STOP-DUB enrolled (1) 237 eligible patients for whom medical treatment had not been successful and who were randomized to either hysterectomy or EA; and (2) an observational cohort of 139 patients who were "provisionally ineligible" or who were eligible but did not wish to be randomized. Enrollment began November 25, 1997 and ended June 30, 2001. Randomized women were followed using telephone interviews at least 2 years and observational women were followed a maximum of 6 months. We also collected information on return clinical center visits and hospital bills from the sites directly. The primary outcome addressed by the randomized trial is the impact of surgery on bleeding, pain, fatigue, and the major problem (symptom) that led the woman to seek treatment for her condition, measured 1 year following surgery. Additional outcomes included the impact of surgery at time points after 1 year; changes in quality of life, activity limitation, sexual functioning, and urinary incontinence; surgical complications; additional surgery; and resource utilization. The costs and the relative cost-effectiveness of the two surgeries will be calculated. The main scientific objective for the observational study was to examine changes over time in terms of treatment selected, DUB-related symptoms, and quality of life. Enrolled women signed an informed consent to participate.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal uterine bleeding in the absence of structural pathology, pharmacologic agents, IUD use, or systemic disorders of hemostasis that could explain the condition.

Exclusion Criteria:

Prescreen

* Age < 18 years
* Postmenopausal status (or bilateral oophorectomy)
* Bleeding not considered excessive by woman
* Desire to retain fertility
* Refusal to consider surgery
* Known myoma (from prior examination)

Eligibility Screen

* Lack of willingness to have a gynecologic or ultrasound examination
* Lack of willingness to be interviewed about bleeding or consider study
* Pregnancy
* Prior endometrial resection or ablation
* Prior myomectomy, myolysis, or hysterectomy

Medical History

* No tentative diagnosis of DUB
* History of malignancy of vagina, cervix, endometrium, or ovary
* History of complex endometrial hyperplasia or simple hyperplasia with atypia
* Current use of tamoxifen
* < 6 months since onset of excessive uterine bleeding
* < 9 months since stopping the use of IUD
* < 9 months since stopping the use of implantable hormone agent
* < 18 months since stopping use of Depo-Provera
* < 6 months of anovulatory DUB after reaching euthyroid status for woman with diagnosis of hypothyroidism
* < 3 months since pathology results indicate presence of endometrial polyp

Baseline Gynecologic Examination

* Enlarged (>= 14 weeks gestational age) uterus
* Focal bleeding of genital, urinary, or gastrointestinal tract

Ultrasound Examination

* Presence of any submucosal myoma
* Presence of any myoma >= 3 cm, any location
* Presence of > 3 myomas, any size or location
* Presence of endometrial polyp(s)
* Malignancy of the vagina, cervix, endometrium, or ovary

Laboratory and Ancillary Tests

* FSH level in women ages > 45 years confirming postmenopausal status
* Abnormal urinary tract or gastrointestinal tract imaging related to uterine bleeding
* Evidence of cervical cancer (screened by Pap smear in last 12 months and confirmed by colposcopy)
* Evidence of complex endometrial hyperplasia or simple hyperplasia with atypia or endometrial cancer (endometrial biopsy in last 12 months)
* Any test value inconsistent with a diagnosis of DUB
* Any test values, unlikely to change, compromising patient safety for surgery

Other

* Any existing medical condition, unlikely to change, putting patient at excessive risk for surgery
* Request for prophylactic bilateral oophorectomy by woman aged <45 years
* Lack of willingness to comply with study requirements
* Uncooperative behavior
* Any coexisting condition that may influence a patient's ability to comply with participation
* Refusal to allow evaluation or follow-up
* In process of scheduling surgery at time of baseline visit

Provisional Eligibility Criteria

* Refusal of randomization
* < 3 months of medical management (excluding GnRH agonist therapy) within the past 2 years
* Ongoing evaluation or treatment for abnormal cervical cytology (including endocervical polyps)
* Gastrointestinal or urinary tract condition unrelated to uterine bleeding currently being treated
* Any temporary test value compromising patient safety
* Any temporary existing medical condition putting patient at excessive risk from surgery
* Any coexisting condition requiring surgery (except tubal occlusion for any woman or oophorectomy for women >= 45 years of age)
* Lack of willingness to proceed with surgery at this time
* Lack of willingness to proceed with surgery likely to result in infertility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242
Dates: Start 1997-11; Study Completion 2004-01

PRIMARY OUTCOMES:
Randomized trial: Impact of surgery on bleeding, pain,
fatigue, and major problem (symptom) leading the woman to seek treatment for her condition.
Observational study: changes over time in treatment selected, DUB-related symptoms, and quality of life.

SECONDARY OUTCOMES:
Randomized trial: Impact of surgery on primary outcomes at time points after 1 year, quality of life, activity limitation, sexual functioning, urinary incontinence, surgical complications, additional surgery, resource utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Kay Dickersin, PhD, Principal Investigator — Brown University

REFERENCES:
- [Background] Dickersin K, Munro M, Langenberg P, Scherer R, Frick KD, Weber AM, Johns A, Peipert JF, Clark M; Surgical Treatments Outcomes Project for Dysfunctional Uterine Bleeding Research Group. Surgical Treatments Outcomes Project for Dysfunctional Uterine Bleeding (STOP-DUB): design and methods. Control Clin Trials. 2003 Oct;24(5):591-609. doi: 10.1016/s0197-2456(03)00023-0. PMID 14500057
- [Background] Weber AM, Munro MG. Endometrial ablation versus hysterectomy: STOP-DUB. Medscape Womens Health. 1998 May;3(3):3. PMID 9732095
- [Derived] Frick KD, Clark MA, Steinwachs DM, Langenberg P, Stovall D, Munro MG, Dickersin K; STOP-DUB Research Group. Financial and quality-of-life burden of dysfunctional uterine bleeding among women agreeing to obtain surgical treatment. Womens Health Issues. 2009 Jan-Feb;19(1):70-8. doi: 10.1016/j.whi.2008.07.002. PMID 19111789
- [Derived] Dickersin K, Munro MG, Clark M, Langenberg P, Scherer R, Frick K, Zhu Q, Hallock L, Nichols J, Yalcinkaya TM; Surgical Treatments Outcomes Project for Dysfunctional Uterine Bleeding (STOP-DUB) Research Group. Hysterectomy compared with endometrial ablation for dysfunctional uterine bleeding: a randomized controlled trial. Obstet Gynecol. 2007 Dec;110(6):1279-89. doi: 10.1097/01.AOG.0000292083.97478.38. PMID 18055721